CLINICAL TRIAL: NCT02617407
Title: Pilot Study -- Oral Microbiome and Dental Plaque Control With Livionex(R) in Children Undergoing Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: Livionex Oral Microbiome and Dental Plaque Control in HSCT Recipients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 15-18297; NCI-2019-00244 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); 160814 (Other: University of California, San Francisco)
Record Dates: First submitted 2015-11-06; First posted 2015-12-01 (Estimated); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Dental Plaque
Keywords: Dental Plaque; Gingivitis; Bacterial Infection; Oral Hygiene; HSCT; Oral Microbiome; Gut Microbiome; Blood Microbiome
MeSH Terms: conditions — Dental Plaque; Gingivitis; Bacterial Infections | interventions — Edetic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Livionex® Dental Gel (Experimental): Study patients assigned to this arm will use Livionex toothpaste for daily teeth brushing from day 1 to day 14. Study participants will be encouraged to continue use study toothpaste and monitored up to 44 days after study enrollment.
  Interventions: Drug: Livionex® Dental Gel; Device: Kolibree Toothbrush
- PreviDent 5000 plus/Tom's of Maine Children's toothpaste (Active Comparator): Study patients assigned to this arm will use PreviDent 5000 plus or Tom's of Maine Children's (age 6 years and younger) toothpaste for daily teeth brushing from day 1 to day 14. Study participants will be encouraged to continue use study toothpaste and monitored up to 44 days after study enrollment.
  Interventions: Drug: PreviDent 5000 plus/Tom's of Maine Children's toothpaste; Device: Kolibree Toothbrush

INTERVENTIONS:
Drug: Livionex® Dental Gel — Oral application Dental Plaque, Gingivitis and Oral Microbiome Control.
  Other Names: Edathamil
  Arms: Livionex® Dental Gel
Drug: PreviDent 5000 plus/Tom's of Maine Children's toothpaste — Oral application for Dental Plaque, Gingivitis and Oral Microbiome Control.
  Other Names: Over the counter toothpaste
  Arms: PreviDent 5000 plus/Tom's of Maine Children's toothpaste
Device: Kolibree Toothbrush — Electric Toothbrush

SUMMARY:
Children undergoing chemotherapy, radiation treatment and Hematopoietic Stem Cell Transplantation (HSCT) have significant difficulties achieving good oral hygiene and dental plaque control. HSCT recipients are at a significant risk for bacteremia and sepsis. Livionex® toothpaste was shown to be effective in reducing dental plaques while containing no additives found in other toothpastes that can cause increased gingival irritation. The investigators hypothesize that improved oral hygiene and better plaque control in pediatric patients receiving chemo/radiation treatment or HSCT may result in reduced oral inflammation, decreased amount of oral bacterial pathogens, and reduced risk of oral-pathogen related systemic bacterial infections. The overall goal of this prospective randomized (2:1) pilot study is to determine whether incorporation of the Livionex® toothpaste in the research regimen could reduce dental plaque.

DETAILED DESCRIPTION:
This is a prospective randomized (2:1) pilot study of children undergoing HSCT or chemo/radiation therapy for cancer treatment who are able to cooperate with saliva collection and dental exams.

RATIONALE:

As chemotherapy and radiation therapy result in a break-down of the mucosal barrier, HSCT recipients and cancer patients are at a significant risk for bacteremia and sepsis from oral pathogens. Children undergoing HSCT have significant difficulties achieving good oral hygiene and dental plaque control because of sensitivity of oral tissues leading to intolerance of teeth brushing and standard dentifrice. This usually results in plaque buildup and moderate to severe gingival inflammation, which persists during and after transplantation. The investigators hypothesize that improved oral hygiene and better plaque control in HSCT recipients and cancer patients may result in reduced oral inflammation, decreased amount of oral bacterial pathogens, and reduced risk of oral-pathogen related bacterial infections.

PRIMARY OBJECTIVES:

To evaluate adherence to oral hygiene by using daily compliance logs and to evaluate the efficacy of Livionex® as compared to standard toothpaste PreviDent® 5000 plus in plaque and gingivitis reduction in HSCT recipients and children receiving chemo/radiation therapy for cancer treatment.

STUDY DURATION:

Therapy 7 days and follow-ups is up to 44 days. It will take 36 months to enroll patients and complete follow-up.

SAFETY ASSESSMENTS:

The incidence of bacteremia with oral pathogens will be followed up to 44 days after first day of intervention. The investigators anticipate that the risk of bacteremia caused by oral pathogens will decrease with study procedures; however, if significantly increased incidence of bacteremia with oral pathogens is documented in either cases or controls, the study will be stopped.

EFFICACY:

The investigators will measure adherence to the protocol of teeth brushing twice per day using test and control dentifrice. The investigators will evaluate the change in dental plaque scores and gingival inflammation from day 0 to 14, and 44 for each patient, as well as compare plaque scores and gingival inflammation between the test and control groups.

At baseline, day 14, and day 44, optical coherence tomography will be used to image and thereby quantify plaque presence. Also, plaque staining will be performed and standardized photographs taken to allow for plaque distribution mapping. On these same days, saliva/dental plaque, stool and blood specimens will be collected to assess for full bacterial profile (microbiome).

UNIQUE ASPECTS:

This study uses a new dentifrice that has been shown to improve plaque control in pediatric cancer patients and HSCT recipients with the goal of improving plaque control during HSCT. This is the first study exploring the composition of plaque and oral microbiome in pediatric HSCT recipients. This study will gather data on the possible link between the oral and gut microbiome with systemic bacteremia during HSCT, the effect of plaque reduction on oral microbiome, and the effect of systemic antibiotic use on oral microbiome.

ELIGIBILITY:
Inclusion Criteria:

* HSCT recipient or chemo/radiation therapy patients who can cooperate with study procedures.
* Parents and patient willing to participate and sign informed consent and assent forms.

Exclusion Criteria:

* Unable to understand or participate in study procedures.
* Known allergy to edathamil or known allergy to multiple hygiene and cosmetic products.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-07-28 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

PRIMARY OUTCOMES:
Adherence to oral hygiene | 7 days
  Compliance will be recorded two times daily, units on a scale 0 - 2 (2 = excellent compliance, 0 = no compliance). A mean score from day 1 to 7 will be compared (t-test) for each patient and between the treatment and the control group.
Plaque index score (Shick R.A., 1961) | 0 to 44 days - change from baseline to day 14 and 44 will be measured
  The following teeth and surfaces will be evaluated for plaque: #A/3 buccal, #E/8 facial, #J/14 buccal, #K/19 lingual, #O/24 facial, and #T/30 lingual. At day 0, 14 and 44 (± 14 days), units on a scale 0 - 3 (0 = absence of dental plaque on the gingival half of the facial surface of a tooth, 1 = the presence of dental plaque covering less than 1/3 of the gingival half of the farcical surface, 2 = the presence of dental plaque covering 1/3 or less than 2/3 of the gingival half of the facial surface, 3 = the presence of dental plaque covering 2/3 or more of the facial surface). A mean score of each time point (day 0, 14, and 44) will be compared (t-test) for each patient longitudinally and between the treatment and the control group.
Gingival index score (Löe H, 1967) | 0 to 44 days - change from baseline to day 14 and 44 will be measured
  The following teeth and surfaces will be evaluated for plaque: #A/3 buccal, #E/8 facial, #J/14 buccal, #K/19 lingual, #O/24 facial, and #T/30 lingual. At day 0, 14 and 44 (± 14 days), units on a scale 0 - 3 (0 = Normal gingiva, 1 = Mild inflammation -- slight change in color, slight edema. No bleeding on probing, 2 = Moderate inflammation-redness, edema and glazing. Bleeding on probing, 3 = Severe inflammation - marked redness and edema. Ulceration. Tendency to spontaneous bleeding). A mean score of each time point (day 0, 14, and 44) will be compared (t-test) for each patient longitudinally and between the treatment and the control group.
Optical Coherence Tomography (OCT) score (Turesky modification of the Quigley-Hein Plaque Index, Ajaharain J, 2014) | 0 to 44 days - change from baseline to day 14 and 44 will be measured
  The following teeth and surfaces will be evaluated for plaque: #A/3 buccal, #E/8 facial, #J/14 buccal, #K/19 lingual, #O/24 facial, and #T/30 lingual. At day 0, 14 and 44 (± 14 days), units on a scale 0 - 5 (0 = No plaque, 1 = Separate flecks of plaque at the cervical margin, 2 = A thin, continuous band of plaque (up to 1 mm) at the cervical margin, 3 = A band of plaque wider than 1 mm, but covering less than 1/3 of the side of the crown of the tooth, 4 = Plaque covering at least 1/3, but less than 2/3 of the side of the crown of the tooth, 5 = Plaque covering 2/3 or more of the side of the crown of the tooth). A mean score of each time point (day 0, 7, and 44) will be compared (t-test) for each patient longitudinally and between the treatment and the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Den Besten, DDS, MS, Principal Investigator — School of Dentistry, UC San Francisco
Locations (1):
- University of California, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No